CLINICAL TRIAL: NCT04223505
Title: Left Atrial Imaging Prior to Cardioversion: Leveraging Computed Tomography to Rule Out Thrombus
Acronym: LACLOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201900117-01H
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEE arm (Active Comparator): TEE will be performed as per clinical routine using multiple standard tomographic planes to rule-out LA/LAA thrombus. Echocardiographic analysis will include: LAA-emptying velocity, and grading the severity of LAA spontaneous ECHO. The severity of the SEC will be graded on a 4 point scale with 1 = minor homogeneous contrast enhancement, 2 = significant homogeneous contrast enhancement, 3 = significant, dense, and inhomogeneous, slow-moving contrast, and 4 = dense slow-moving contrast.
  Interventions: Diagnostic Test: Transesophageal Echocardiography (TEE)
- CCT arm (Experimental): As per local protocol, a non-contrast enhanced prospective ECG-triggered image acquisition will be acquired. This will be followed by a contrast-enhanced prospective ECG-triggered will be acquired using a tri-phasic contrast protocols. Delayed CT images will be acquired 60 seconds after the initial contrast-enhanced CT scan.Cardiac CT image interpretation will be performed as per clinical routine. The LA and LAA will be assess for filling defects and characterized based upon attenuation values. If LA/LAA thrombus cannot be excluded, filling defects will be assessed on the delay images. Increases in attenuation would be consistent with pseudo-thrombus from 'slow flow' and 'incomplete opacification'. Areas where attenuation does not change significantly (persistent filling defect) will be diagnosed as thrombus. It will be recommended that patients with thrombus will undergo TEE.
  Interventions: Diagnostic Test: Contrast enhanced ECG-gated cardiac CT (CCT); Diagnostic Test: Transesophageal Echocardiography (TEE)

INTERVENTIONS:
Diagnostic Test: Contrast enhanced ECG-gated cardiac CT (CCT) — Contrast enhanced ECG-gated cardiac CT (CCT) is a sensitive, noninvasive alternative method used to exclude of left atrial and LAA thrombus. CCT provides high spatial and good temporal resolution and its ability to detect thrombus has been evaluated. CCT, compared to TEE, for the exclusion of thrombus in the LAA had a sensitivity and specificity of 100% and 99.3%, respectively. A high sensitivity is needed to minimize risk of embolus, and if a thrombus is detected on CT, a confirmatory TEE may be performed or patients may receive anticoagulation. Some argue that the potential benefits of CT and its lower associated procedural risk, the risk:benefit ratio would still favour CT.
  Arms: CCT arm
Diagnostic Test: Transesophageal Echocardiography (TEE) — TEE is considered the reference standard to rule-out left atrial (LA) and left atrial appendage (LAA) thrombus prior to cardioversion. Several studies have examined the accuracy of TEE for detecting LAA thrombus. Compared to autopsy and intraoperative findings, TEE has a mean sensitivity of 100% and mean specificity of 99%. Although the gold standard, a TEE-guided therapy is still associated with an embolic rate of 0.8%.

SUMMARY:
Evaluating contrast enhanced ECG-gated cardiac CT (CCT) as an alternative to transesophageal echocardiography (TEE) to expedite cardioversion of atrial fibrillation (AF), improve patient care and reduce hospital admissions for AF and atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted patients who require LA imaging prior to cardioversion
2. Age ≥18 years old
3. Able and willing to comply with the study procedures

Exclusion Criteria:

1. Indication for acute cardioversion (e.g. hemodynamic instability, acute coronary syndrome (ACS), or pulmonary edema)
2. Unwillingness or inability to provide informed consent
3. Contraindication to Cardiac CT

   * Severe renal insufficiency(GFR< 45ml/min)
   * Allergy to intravenous contrast agents
   * Contraindications to radiation exposure (for example, pregnancy)
   * Inability to perform 20-second breath-hold
4. Contraindication to TEE

   * Unrepaired tracheoesophageal fistula
   * Esophageal obstruction or stricture
   * Perforated hollow viscus
   * Poor airway control
   * Severe respiratory depression
   * Uncooperative, unsedated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD, Principal Investigator — UOHI
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 102 participants, 52 were randomized to CCT and 50 to TEE
Groups:
- CCT Arm: A non-contrast enhanced prospective ECG-triggered image acquisition will be acquired. This will be followed by a contrast-enhanced prospective ECG-triggered will be acquired using tri-phasic contrast protocols. Delayed CT images will be acquired 60 seconds after initial contrast-enhanced CT scan.Cardiac CT image interpretation will be performed as per clinical routine. The LA and LAA will be assess for filling defects and characterized based upon attenuation values. If LA/LAA thrombus cannot be excluded, filling defects will be assessed on the delay images. Increases in attenuation would be consistent with pseudo-thrombus from 'slow flow' and 'incomplete opacification'. Areas where attenuation does not change significantly (persistent filling defect) will be diagnosed as thrombus. It will be recommended that patients with thrombus will undergo TEE.
  Contrast enhanced ECG-gated cardiac CT (CCT): Contrast enhanced ECG-gated cardiac CT (CCT) is a sensitive, noninvasive alternative method used to exclude left atrial and LAA thrombus. CCT provides high spatial and good temporal resolution and its ability to detect thrombus has been evaluated.
Period: Overall Study
Arm/Group | TEE Arm | CCT Arm
Started | 50 | 52
Completed | 42 | 52
Not Completed | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEE Arm | CCT Arm | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.8) | 66.3 (11.3) | 66.76 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 36 | 38 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Time to Imaging
Description: This outcome was measured by calculating the time between admission and imaging.
Time Frame: From admission to imaging/spontaneous cardioversion, up to approximately 30 days.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TEE Arm | CCT Arm
Number analyzed (Participants) | 50 | 52
hours | 28.1 (34.9) | 7.1 (12.5)

2. Secondary Outcome: Time to Cardioversion
Description: This outcome was measured by calculating the time between admission and cardioversion.
Time Frame: From admission to cardioversion, up to approximately 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEE Arm | CCT Arm
Number analyzed (Participants) | 50 | 52
days | 4.6 (11.1) | 1.7 (1.8)

3. Other Pre Specified Outcome: Time to Hospital Discharge
Description: This outcome was measured by calculating the time between admission and hospital discharge.
Time Frame: From admission to hospital discharge, up to approximately 90 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TEE Arm | CCT Arm
Number analyzed (Participants) | 50 | 52
days | 6.7 (6.9) | 7.0 (10.8)

4. Other Pre Specified Outcome: QoL
Description: This outcome was calculated from the following QoLs: European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) and Atrial Fibrillation Impact (AFImpact). EQ-5D-5L health score is a continuous scale from 0 to 100 with 100 being the best outcome. AFImpact scores were calculated using a seven-point Likert Scale (1=none of the time, 7=all of the time). AFImpact-Vitality, Emotional Distress, Sleep score (AFImpact-VEDS) was calculated using all questions in the questionnaire. The difference between AFImpact-VEDS scores at hospital admission and discharge was calculated where minimum change in score is 0 and maximum change in score is 108. AFImpact-emotional distress subscale score was calculated using 8 questions about emotional distress. The difference between AFImpact emotional distress scores at hospital admission and discharge was calculated where minimum change in score is 0 and maximum change in score is 48. The higher change in AFImpact scores represented a better outcome.
Time Frame: At hospital discharge
Measure: Mean (Standard Deviation); unit: score
Arm/Group | TEE Arm | CCT Arm
Number analyzed (Participants) | 50 | 52
score
  European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | 68.1 (18.2) | 75.3 (15.5)
  AFImpact-Vitality, Emotional Distress, Sleep score (AFImpact-VEDS) | 8.5 (4.2) | 7.5 (3.5)
  Atrial Fibrillation Impact (AFImpact)-emotional distress | 3.0 (1.8) | 2.4 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 months.
Arm/Group | TEE Arm | CCT Arm
All-Cause Mortality (participants affected / at risk) | 1/50 | 1/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 14/50 | 17/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEE Arm (N=50) | CCT Arm (N=52)
Renal impairment (Renal and urinary disorders) | 14 | 17 — 25% increase in baseline creatinine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT04223505/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04223505/ICF_001.pdf